CLINICAL TRIAL: NCT06268938
Title: Outcomes of Mastoid Obliteration Canal Wall Down Tympanomastoidectomy in Cholesteatoma Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Abdelal Mohamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mastoid obliteration
Record Dates: First submitted 2023-11-27; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cholesteatoma
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle obliteration (Experimental): Mastoid cavity obliteration by muscle
  Interventions: Procedure: Canal wall down tympanomastoidectomy
- Bone obliteration (Active Comparator): Mastoid cavity obliteration by bone
  Interventions: Procedure: Canal wall down tympanomastoidectomy

INTERVENTIONS:
Procedure: Canal wall down tympanomastoidectomy — Mastoid cavity obliteration by in canal wall down tympanomastoidectomy tympanomastoidectomy in cholesteatoma surgery

SUMMARY:
Randomised study to evaluate the outcomes of mastoid cavity obliteration by muscle versus bone in canal wall down tympanomastoidectomy in cholesteatoma surgery

DETAILED DESCRIPTION:
Regarding discharge Time of epithelizqtion Hearing outcomes Quality of life

ELIGIBILITY:
Inclusion Criteria:

* all patients who have extensive or recuutrent cholesteatoma undergoing canal wall down tympanomastoidectomy

Exclusion Criteria:

* not willing for surgery
* Malignancy

  * Patients with intracranial complication
* Residual cholesteatoma

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Size of mastoid cavity in mm | 1 month
  Endoscopic examination of the mastoid cavity after 1month to evaluate the degree of epithelization and if there is discharge .

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut university hospital, Asyut
  - Rehab Abd Elal Mohammed, Asyut

REFERENCES:
- [Background] Mehta RP, Harris JP. Mastoid obliteration. Otolaryngol Clin North Am. 2006 Dec;39(6):1129-42. doi: 10.1016/j.otc.2006.08.007. PMID 17097437
- [Background] Khalil HS, Windle-Taylor PC. Canal wall down mastoidectomy: A long term commitment to the outpatients? BMC Ear Nose Throat Disord. 2003 Sep 4;3(1):1. doi: 10.1186/1472-6815-3-1. PMID 12956889
- [Background] Illes K, Meznerics FA, Dembrovszky F, Fehervari P, Banvolgyi A, Csupor D, Hegyi P, Horvath T. Mastoid Obliteration Decreases the Recurrent and Residual Disease: Systematic Review and Meta-analysis. Laryngoscope. 2023 Jun;133(6):1297-1305. doi: 10.1002/lary.30413. Epub 2022 Sep 28. PMID 36169349
- [Background] Krol B, Cywka KB, Skarzynska MB, Skarzynski PH. Mastoid obliteration with S53P4 bioactive glass after canal wall down mastoidectomy: Preliminary results. Am J Otolaryngol. 2021 Mar-Apr;42(2):102895. doi: 10.1016/j.amjoto.2020.102895. Epub 2021 Jan 5. PMID 33429176
- [Background] Weiss NM, Bachinger D, Botzen J, Grossmann W, Mlynski R. Mastoid cavity obliteration leads to a clinically significant improvement in health-related quality of life. Eur Arch Otorhinolaryngol. 2020 Jun;277(6):1637-1643. doi: 10.1007/s00405-020-05881-4. Epub 2020 Mar 6. PMID 32144569